CLINICAL TRIAL: NCT07145983
Title: Peer Support Intervention Effect on Medication Adherence, Self-care and Knowledge Among Patients With Diabetes: A Randomized Control Trial
Brief Title: Effect of Peer Support Intervention on Medication Adherence, Self-care and Knowledge Among Patients With Diabetes
Acronym: DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Collaborators: Mekelle University (Other)
Responsible Party: Principal Investigator, Halefom Kahsay Haile, Mr, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Addis Ababa University(AAU); 084/24/SoP (Other: Addis Ababa University)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Peer Influence; Medication Adherence; Self Care
Keywords: Diabetes Mullites; Peer support; Medication adherence; self-care Practice; Diabetes Knowledge
MeSH Terms: conditions — Medication Adherence | interventions — Self Care; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive peer-led support sessions in addition to usual diabetes care.
  Interventions: Behavioral: Structured Diabetes Education on medication Adherence and self care
- No-Intervention Comparator: Standard Care Alone(Control group) (No Intervention): Participants continue with routine follow-up and standard diabetes care only.

INTERVENTIONS:
Behavioral: Structured Diabetes Education on medication Adherence and self care — Lived-experience facilitation, goal setting, real-world problem solving, and ongoing peer accountability not provided in standard clinician-led education. Peer-led, group-based sessions emphasizing lived experiences, problem-solving, and mutual support. Participants meet regularly in small groups facilitated by trained peers with diabetes. Includes structured booster follow-ups and SMS reminders to reinforce adherence and self-care.
  Other Names: Structured Diabetes Education on Diabetes definition, sign and symptoms and management
  Arms: Intervention Group

SUMMARY:
The goal of this interventional study is to learn about the effect of a peer support group intervention on adherence, self-care practice, and knowledge among diabetic patients on follow-up care. The main question it aims to answer is:

* Does participation in a peer support group improve medication adherence, self-care behaviors, and diabetes knowledge compared to standard care?
* Participants with diabetes who are already receiving follow-up care at Ayder Comprehensive Specialized Hospital will be randomly assigned to either a peer support group (intervention group) or continue their usual follow-up care (control group). Outcomes will be measured through validated questionnaires and pill counts over the study period.

DETAILED DESCRIPTION:
BACKGROUND Diabetes mellitus (DM) is a chronic metabolic disorder that comes as one of the fastest-growing global health challenges, with the number of affected individuals projected to reach 643 million by 2030 and 783 million by 2045. Sub-Saharan Africa is experiencing a rapid rise in DM prevalence, partly due to urbanization, lifestyle changes, and limited access to preventive and treatment services. In Ethiopia, diabetes contributes substantially to the burden of non-communicable diseases, yet many patients fail to achieve optimal glycemic control.

Peer support is considered a promising, feasible, and culturally appropriate enhancement to diabetes care, enabling participants to assist one another in their ongoing self-management efforts. It is effective in preventing the complications of diabetes and enhancing health outcomes in patients with diabetes. Previous systematic reviews have reported that programs were effective for diabetes outcomes, including glycemic control, knowledge of diabetes, self-management skills, and self-efficacy. A healthy lifestyle, an appropriate diet, and medication adherence among diabetic patients are essential factors in the prevention of diabetes complications as well as maintaining good glycemic control. However, many patients with diabetes fail to manage the disease due to its complex nature. Hence, patients with diabetes need self-management education to assist them in comprehending and dealing with the disease.

Several rigorous reviews have demonstrated that adherence to treatment among patients with chronic diseases in developed countries is about 50%. Considering the scarcity and inequities in access to healthcare services in developing countries, this rate is assumed to be even lower. Poor adherence to diabetes medications is common among African Americans and contributes to these disproportionally worse outcomes. Numerous studies suggested that diabetic peer support programs have positive outcomes on improvement of adherence to medication which is essential for successful diabetes management. For example, Shiyanbola and coworker supported that conduction of an efficacy trial to address medication adherence using a peer-supported tailored intervention is essential. The healthcare effectiveness report from USA point out that inadequate medication adherence is one of the main causes of the differences in glycemic control attainment rates between real-world settings and randomized controlled trials which emphasize the need for better provider and patient support programs to improve adherence.Thus, Patient support programs can improve persistence with and/or adherence to medications for the treatment of chronic diseases like diabetes.

Sub-Saharan Africa researches have demonstrated that peer support programs are beneficial and enabling participants to modify their lifestyle and adhere to treatment. A study conducted in Uganda showed that improvements in eating habits, diastolic blood pressure, and glycosylated hemoglobin (A1C), after peer support program had carried out to diabetic patients and concluded that as it is a workable intervention to enhance diabetes care in health care settings. Additionally, diabetes peer support programs have been demonstrated to enhance patients' health-related behaviors, metabolic management, and quality of life in nations such as South Africa, and Cameroon. After the diabetes peer support program has positively impacted its members in Malawi, the researchers suggested that additional recruitment and ongoing training for peer supporters is necessary to reinforce and update management knowledge and skills. Besides, they concluded that it is a viable strategy for the non-communicable diseases unit within the Ministry of Health. In Ethiopia, fewer than 50% of diabetic individuals obtain proper diabetes care.

Despite the empirical studies showing positive and significant relationships between diabetes peer support and treatment adherence among patients with diabetes, the exact mechanism by which peer support affects patient adherence is not yet completely understood. Further research is needed to address how the differences in types of support, such as functional or emotional support, are linked to outcomes for patients. Specifically, there remains a gap in understanding what constitutes peer support and how to effectively implement it in low-resource environments, like Ethiopia health care settings.

Patient education materials provided by diabetes focused organizations do not increase patient self efficacy or engagement with self management as these documents contain complex medical jargon and provide only general guidelines, not patient-specific instruction. Peer support interventions, where individuals with lived experience of diabetes share advice, encouragement, and practical strategies, offer a potentially powerful extension of these existing support systems. Such programs have demonstrated benefits in enhancing treatment adherence, self-care practices, and disease-related knowledge in various settings. Despite this, there is limited data from Ethiopia on the effect of structured peer support groups among patients receiving care in tertiary hospitals.

This study assesses the effectiveness of a structured peer support group in enhancing medication adherence, self-care behaviors, and diabetes-related knowledge among adult patients attending follow-up at Ayder Comprehensive Specialized Hospital, a tertiary care facility in northern Ethiopia. The findings aim to inform efforts to integrate peer support into routine diabetes care within similar low-resource environments.

METHODOLOGY and MATERIALS Study Setting The study was conducted at Ayder Comprehensive Specialized Hospital (ACSH), the largest referral hospital in the Tigray region, situated in Mekelle city, about 780 kilometers north of Addis Ababa, Ethiopia's capital. ACSH serves an estimated 10 million people from Tigray and neighboring regions, including Amhara and Afar. With a capacity of 500 beds, the hospital manages approximately 10,000 inpatient admissions and 100,000 outpatient visits annually.

The diabetic clinic at ACSH is a major center for diabetes management, providing follow-up care for around 5,000 patients. Outpatient services are delivered two days a week, serving more than 100 patients per visit. The clinic is operated by two Senior physicians, residents and five nurses who provide a range of essential services, such as diabetes education, individualized counseling on diet, emergency care, medication adherence, and insulin administration. Antidiabetic treatments are adjusted based on fasting blood glucose and HbA1C results. Newly diagnosed patients receive intensive follow-up during the first six months to help maintain optimal blood glucose levels.

Study Design and Period A randomized controlled trial (RCT) design was employed from January to September 2025 to evaluate the effect of a peer support intervention among patients with diabetes attending Ayder Comprehensive Specialized Hospital (ACSH).

Study Population The study involved diabetic patients aged 18 to 65 years who were receiving follow-up care at ACSH. Participants were divided into three groups whose were categorized as the peer support group, the intervention group and the control group. Eligible participants of the peer support group had a minimum of 10th grade educational background with more than three years of disease duration, stable glycemic control, a documented history of regular follow-up at ACSH. Besides, the intervention group were those who received the peer-led educational sessions, which aimed to improve adherence to diabetes treatment, enhance self-care behaviors, and increase diabetes-related knowledge.

Sample Size Determination The sample size for this study was determined separately for the peer support group and the two comparison groups. Five participants were purposively selected for the peer support group based on predefined eligibility criteria. Selection was done in collaboration with clinical service providers at the diabetic center to ensure the inclusion of experienced individuals, following guidance from validated studies on peer support interventions for diabetic patients. For the intervention and control groups, the sample size was calculated using the statistical superiority design formula for continuous variables: n = [(Z₁ + Z₂)² × (2S²)] / d². In this formula, Z₁ represents the z-score for a 95% confidence level (1.96), Z₂ corresponds to a power of 80% (0.84). The standard deviation (S = 4) was estimated based on the range of scores from the Morisky Medication Adherence Scale with eight items (MMAS-8), which spans from 0 (indicating poor adherence) to 8 (indicating high adherence). A minimum clinically meaningful difference of 2 points (d = 2) in adherence scores between the groups was considered for sample size calculation. This calculation provided the required sample size for the intervention and control groups to detect a meaningful difference in adherence outcomes. A total of 100 eligible patients with diabetes were recruited using a simple random sampling method with 50 participants assigned to the intervention group and 50 to the control group.

Standard Care Scheduled consultations with a physician, laboratory investigations and medication refill were the standard care services delivered for patients with diabetes during the clinic's service days at the diabetic center of the Hospital. Follow-up appointments are typically scheduled every two to three months. Newly diagnosed patients receive individualized counseling from the nurse on duty, addressing diabetes-related and patient-specific concerns. Additionally, patients collect their prescribed medications from the hospital pharmacy up on visiting the hospital for follow up in which standard pharmacy care had also served. Thus, in this trial both groups were received this standard health care service equally.

Peer Support Intervention and Procedures The study was conducted in two phases. Phase I involved the recruitment and preparation of the peer support group (n = 5), which took place from October to November 2024. These individuals were selected in advance and remained consistent throughout the intervention period. One registered nurse was recruited to serve as a facilitator for the peer support sessions. A two-day training was provided to the peer supporters by the principal investigator (PI) and the facilitator which included role-playing exercises to prepare them for effective communication and engagement with intervention group members. They were primarily trained to educate and share their experience to peers on scheduled sessions focused on treatment adherence, self-care behaviors, and diabetes-related knowledges.

On Phase II, enrollment of the intervention and control group was continued during their regular appointments at the diabetic clinic. Both groups were matched in terms of sociodemographic characteristics and disease-related factors. While the control group received baseline assessments only and continued with standard care, members of the intervention group attended a one-hour orientation session to explain the study's objectives, potential risks of withdrawal, and the importance of sustained participation. Following this, each peer supporter was assigned to a group of 10 intervention participants, forming five peer-led support groups.

The peer support intervention was delivered through scheduled. It was a one-hour group session which arranged with the regular clinic appointments and conducted for three rounds every two months (at 2,4 and 6 month) over the study period for each group. Each group member was expected to participate in all the three sessions, which were structured around three core components: (a) sharing personal experiences and knowledge about diabetes and its complications, blood glucose triggering factors and providing psychosocial support focused on the self-management (disease-related component); (b) offering education and encouragement for medication adherence (medication adherence component); and (c) supporting the integration of dietary and physical activity recommendations into daily routines (behavioral component). All group sessions were audio-recorded and reviewed to assess adherence to the intervention protocol. Additionally, the principal investigator conducted weekly follow-up phone calls with the peer supporters to document the topics covered during each session and address any challenges encountered during the implementation. Monthly debriefing sessions were conducted to discuss their experiences and challenges. Feedback on their performance was provided based on audio recordings of the group sessions.

Data collection Instruments and Measurements Data were collected using participant interviews, review of medical records as well as adapted diabetes questionnaires for each outcome variable in the intervention and control groups. Four clinical pharmacists were recruited to collect the consecutive data whose were not aware of the group to which the respondent belongs.

Data Analysis Data were entered into EpiData version 4.6 and exported to SPSS version 25 for analysis. Descriptive statistics such as frequencies, percentages, means, and standard deviations were used to summarize sociodemographic, clinical, and behavioral characteristics of participants. Medication adherence, diabetes knowledge, and self-care practice scores were calculated according to their respective validated scales. The effect of the peer support group intervention within-group and between-group was assessed and comparisons were performed. Paired t-tests were used to determine changes in the outcome variables within each group (intervention and control) before and after the intervention. Independent sample t-tests were applied to compare mean differences between groups. Furthermore, a Difference-in-Differences (DiD) approach was employed to evaluate the net effect of the intervention by comparing the changes in outcomes from baseline to follow-up between the intervention and control groups. Bivariate logistic regression was first conducted to explore associations between independent variables and outcome measures. Variables with a p-value < 0.25 were entered into multivariable logistic regression to control for potential confounders. Adjusted odds ratios (AOR) with 95% confidence intervals (CI) were reported, and statistical significance was set at p < 0.05. Model adequacy was verified using the Hosmer-Lemeshow goodness-of-fit test.

RESULT (In Progress)

ELIGIBILITY:
Inclusion Criteria:

* Clincal Diagnosis of Diebetes mullites's Disease
* Must be on at least one diabetes medication
* Must had at least two concicative follow-up visits at the Diabetes clinic

Exclusion Criteria:

* Declined to participate in any of the group
* Concurrent endocrine disorders (thyroid disease, obesity, or gestational diabetes)
* Chronic diseases (cardiac heart failure, hepatitis and cancer)
* Enrollement in other educational programs during the study period those who
* Health professionals with diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Medication Adherence status | Baseline and 6 months
  Medication adherence of each group was assessed through a mixed method using the Morisky Medication Adherence Scale (MMAS-8) and self-reported pill count. The Morisky Medication Adherence Scale consisted of seven dichotomous items and one item rated on a five-point Likert scale which provided five response options, scored from 0 to 1 in 0.25-point increments. Based on the total score, patients were classified as low adherers (score <6), medium adherers (score 6 to <8),or high adherers (score = 8). Pill count data were obtained at each assessment round to evaluate actual medication use. Adherence was calculated by subtracting the number of pills remaining from the quantity dispensed, dividing the result by the product of the prescribed daily dose and the number of days since the last refill, and then multiplying by 100 to obtain a percentage. Patients with adherence below 80% were classified as Poor adherent, and those with above 80% were classified as Good adherent.
Self care Practice Status | Baseline and 6 months
  Self-care practices were measured using the Summary of Diabetes Self-Care Activities (SDSCA) scale, which captures partcipants previous seven days self care activties of the five key domains(Diet,Exercise, blood-glucose testing,foot-care and compliance to recommended treatmens).The Difference in mean score of each dommain was used to compare between groups.
Knowlege status on Diabetes | Baseline and 6 months
  Diabetes-related knowledge was assessed using a structured questionnaire adapted from the Diabetes Knowledge Test (DKT). The instrument included 14 core items administered to all participants, with an additional 9 items for insulin users. Each correct response was scored as 1, and incorrect or "don't know" responses were scored as 0. Non-insulin users were scored out of 14 points, while insulin users were scored out of 23 points. Participants were classified as having good knowledge if their score exceeded the mean, and poor knowledge if their score was at or below the mean.

SECONDARY OUTCOMES:
Factors associated with Medication adherence,selfcar prectics and knowledg of Diabetes | 6 months
  Bivariant and Multiple regression analysis was done to determine significant factors associted with the primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Halefom K Haile, Msc, Principal Investigator — Addis Ababa University, Adigrat university; Teferi G Fenta, Professor, Study Chair — Addis Ababa University; Bruck M Habte, PhD, Study Director — Addis Ababa University
Locations (1):
- Ayder Comprehensive Specialized Hospital (Mekelle University Hospital), Mek'ele, Tigray, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Currently, our data needs clearance,organization and documentation

REFERENCES:
- [Background] Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF DIABETES ATLAS [Internet]. 10th edition. Brussels: International Diabetes Federation; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK581934/ PMID 35914061
- [Background] Atun R, Davies JI, Gale EAM, Barnighausen T, Beran D, Kengne AP, Levitt NS, Mangugu FW, Nyirenda MJ, Ogle GD, Ramaiya K, Sewankambo NK, Sobngwi E, Tesfaye S, Yudkin JS, Basu S, Bommer C, Heesemann E, Manne-Goehler J, Postolovska I, Sagalova V, Vollmer S, Abbas ZG, Ammon B, Angamo MT, Annamreddi A, Awasthi A, Besancon S, Bhadriraju S, Binagwaho A, Burgess PI, Burton MJ, Chai J, Chilunga FP, Chipendo P, Conn A, Joel DR, Eagan AW, Gishoma C, Ho J, Jong S, Kakarmath SS, Khan Y, Kharel R, Kyle MA, Lee SC, Lichtman A, Malm CP, Mbaye MN, Muhimpundu MA, Mwagomba BM, Mwangi KJ, Nair M, Niyonsenga SP, Njuguna B, Okafor OLO, Okunade O, Park PH, Pastakia SD, Pekny C, Reja A, Rotimi CN, Rwunganira S, Sando D, Sarriera G, Sharma A, Sidibe A, Siraj ES, Syed AS, Van Acker K, Werfalli M. Diabetes in sub-Saharan Africa: from clinical care to health policy. Lancet Diabetes Endocrinol. 2017 Aug;5(8):622-667. doi: 10.1016/S2213-8587(17)30181-X. Epub 2017 Jul 5. No abstract available. PMID 28688818
- [Background] Gebreyohannes EA, Netere AK, Belachew SA. Glycemic control among diabetic patients in Ethiopia: A systematic review and meta-analysis. PLoS One. 2019 Aug 27;14(8):e0221790. doi: 10.1371/journal.pone.0221790. eCollection 2019. PMID 31454396
- [Background] Fisher EB, Boothroyd RI, Elstad EA, Hays L, Henes A, Maslow GR, Velicer C. Peer support of complex health behaviors in prevention and disease management with special reference to diabetes: systematic reviews. Clin Diabetes Endocrinol. 2017 May 25;3:4. doi: 10.1186/s40842-017-0042-3. eCollection 2017. PMID 28702258
- [Background] Funnell MM. Peer-based behavioural strategies to improve chronic disease self-management and clinical outcomes: evidence, logistics, evaluation considerations and needs for future research. Fam Pract. 2010 Jun;27 Suppl 1(Suppl 1):i17-22. doi: 10.1093/fampra/cmp027. Epub 2009 Jun 9. PMID 19509083
- [Background] Azmiardi A, Murti B, Febrinasari RP, Tamtomo DG. The effect of peer support in diabetes self-management education on glycemic control in patients with type 2 diabetes: a systematic review and meta-analysis. Epidemiol Health. 2021;43:e2021090. doi: 10.4178/epih.e2021090. Epub 2021 Oct 22. PMID 34696569
- [Background] Gutierrez AP, Fortmann AL, Savin K, Clark TL, Gallo LC. Effectiveness of Diabetes Self-Management Education Programs for US Latinos at Improving Emotional Distress: A Systematic Review. Diabetes Educ. 2019 Feb;45(1):13-33. doi: 10.1177/0145721718819451. Epub 2018 Dec 20. PMID 30569831
- [Background] Debussche X, Besancon S, Balcou-Debussche M, Ferdynus C, Delisle H, Huiart L, Sidibe AT. Structured peer-led diabetes self-management and support in a low-income country: The ST2EP randomised controlled trial in Mali. PLoS One. 2018 Jan 22;13(1):e0191262. doi: 10.1371/journal.pone.0191262. eCollection 2018. PMID 29357380
- [Background] Khare J, Jindal S. Observational study on Effect of Lock Down due to COVID 19 on glycemic control in patients with Diabetes: Experience from Central India. Diabetes Metab Syndr. 2020 Nov-Dec;14(6):1571-1574. doi: 10.1016/j.dsx.2020.08.012. Epub 2020 Aug 20. PMID 32858474
- [Background] Lee AA, Piette JD, Heisler M, Janevic MR, Rosland AM. Diabetes self-management and glycemic control: The role of autonomy support from informal health supporters. Health Psychol. 2019 Feb;38(2):122-132. doi: 10.1037/hea0000710. PMID 30652911
- [Background] Shiyanbola OO, Maurer M, Mott M, Schwerer L, Sarkarati N, Sharp LK, Ward E. A feasibility pilot trial of a peer-support educational behavioral intervention to improve diabetes medication adherence in African Americans. Pilot Feasibility Stud. 2022 Nov 14;8(1):240. doi: 10.1186/s40814-022-01198-7. PMID 36376960
- [Background] Edelman SV, Polonsky WH. Type 2 Diabetes in the Real World: The Elusive Nature of Glycemic Control. Diabetes Care. 2017 Nov;40(11):1425-1432. doi: 10.2337/dc16-1974. Epub 2017 Aug 11. PMID 28801473
- [Background] Burudpakdee C, Khan ZM, Gala S, Nanavaty M, Kaura S. Impact of patient programs on adherence and persistence in inflammatory and immunologic diseases: a meta-analysis. Patient Prefer Adherence. 2015 Mar 11;9:435-48. doi: 10.2147/PPA.S77053. eCollection 2015. PMID 25792817
- [Background] Zachariah R, Teck R, Buhendwa L, Fitzerland M, Labana S, Chinji C, Humblet P, Harries AD. Community support is associated with better antiretroviral treatment outcomes in a resource-limited rural district in Malawi. Trans R Soc Trop Med Hyg. 2007 Jan;101(1):79-84. doi: 10.1016/j.trstmh.2006.05.010. Epub 2006 Sep 8. PMID 16962622
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Fitzgerald JT, Funnell MM, Hess GE, Barr PA, Anderson RM, Hiss RG, Davis WK. The reliability and validity of a brief diabetes knowledge test. Diabetes Care. 1998 May;21(5):706-10. doi: 10.2337/diacare.21.5.706. PMID 9589228
- See also: World Health Organization. Adherence to long-term therapies: evidence for action. — http://apps.who.int/medicinedocs/en/d/Js4883e/.2003.
- See also: Book chapter on assessing diabetes self-management summary diabetes self-care activities questionnaire — https://www.taylorfrancis.com/chapters/edit/10.4324/9781315077369-20/assessing-diabetes-self-management-summary-diabetes-self-care-activities-questionnaire-deborah-toobert-russell-glasgow